CLINICAL TRIAL: NCT01484938
Title: Lens Wearing Experience and Biocompatibility of a Marketed Multi-Purpose Disinfecting Solution in Silicone Hydrogel and Soft Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C-10-017
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Results first posted 2012-10-08 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Refractive Error
Keywords: Soft contact lenses; Multi-purpose solution; Corneal staining
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPTI-FREE (Experimental): OPTI-FREE PureMoist multi-purpose contact lens solution used for cleaning, rinsing, disinfecting/storing, and reinserting contact lenses, per protocol-specified regimen
  Interventions: Device: OPTI-FREE PureMoist

INTERVENTIONS:
Device: OPTI-FREE PureMoist — Commercially marketed multi-purpose contact lens solution for cleaning, rinsing, disinfecting/storing, and reinserting contact lenses

SUMMARY:
The purpose of this study was to describe mean differences in corneal staining (type and area) for OPTI-FREE PureMoist Multi-Purpose Disinfecting Solution (MPDS) at Day 30 compared to Baseline (Day 0).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Soft contact lens wear on a daily wear basis
* Able to wear contact lenses for at least 8 hours
* Generally healthy and have normal ocular health
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* No use of additional lens cleaners
* No known sensitivities to any ingredient in the test article
* No history of ocular surgery/trauma within the last six months
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jami R Kern, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 study centers in the Netherlands, 3 study centers in Sweden, and 1 study center in Australia.
Groups:
- OPTI-FREE: Multi-purpose contact lens solution used for cleaning, rinsing, disinfecting/storing, and reinserting contact lenses, per protocol-specified regimen.
Period: Overall Study
Arm/Group | OPTI-FREE
Started | 175
Completed | 171
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — Noncompliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | OPTI-FREE
Number analyzed (Participants) | 175
Age Continuous [Mean (Standard Deviation); unit: years] | 37.6 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 64
Region of Enrollment [Number; unit: participants]
  Netherlands | 72
  Sweden | 75
  Australia | 28

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Day 0) in Average Corneal Staining Area at Day 30
Description: Percentage corneal staining was assessed by the investigator for each of five regions of the cornea; i.e., four quadrants plus central. The investigator instilled flourescein dye and examined the cornea with a slit lamp, i.e., biomicroscope and yellow filter. Percentage corneal staining was recorded in increments of ten, and the percentages of the five regions were averaged together.
Time Frame: Baseline (Day 0), Day 30
Population: Intent to treat. All subjects who were enrolled in the study and completed at least one on-regimen study visit were evaluable for intent-to-treat analyses.
Measure: Mean (Standard Deviation); unit: Percentage of corneal staining
Arm/Group | OPTI-FREE
Number analyzed (Participants) | 171
Percentage of corneal staining | -5.04 (16.119)

2. Primary Outcome: Mean Change From Baseline (Day 0) in Total Corneal Staining Type at Day 30
Description: Corneal staining type was assessed by the investigator for each of five regions of the cornea, i.e., four quadrants plus central. The investigator instilled flourescein dye and examined the cornea with a slit lamp, i.e., biomicroscope and yellow filter. Corneal staining type was recorded on a 5-point scale for each region: 0=none; 1=micropunctate; 2=macropunctate; 3=coalesced macropunctate; 4=patch (>/= 1 mm). The five regions were summed, for a summed total range of 0-20.
Time Frame: Baseline (Day 0), Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPTI-FREE
Number analyzed (Participants) | 171
Units on a scale | -0.82 (1.777)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 3 months, 2 weeks, 2 days.
Description: All subjects enrolled in the study and exposed to test regimen were evaluable for safety analyses.
Arm/Group | OPTI-FREE
Serious Adverse Events (participants affected / at risk) | 0/175
Other Adverse Events (participants affected / at risk) | 0/175

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.